CLINICAL TRIAL: NCT04749251
Title: IDEAL Blood Pressure Management During Endovascular Therapy for Acute Ischemic Stroke:A Feasibility Study of Randomisation to Individual vs. Fixed Blood Pressure Targets During Endovascular Therapy for Acute Ischemic Stroke
Brief Title: IDEAL Blood Pressure Management During Endovascular Therapy for Acute Ischemic Stroke
Acronym: IDEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg University (Other); Klinikum Kassel (Other); University Hospital Heidelberg (Other); Sahlgrenska University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IDEAL BP Feasibility Study
Record Dates: First submitted 2021-01-29; First posted 2021-02-11 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2021-01

CONDITIONS: Acute Ischemic Stroke
Keywords: Endovascular therapy; Blood pressure; Anesthesia
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: The study will be performed as a single center study, conducted at Aarhus University Hospital, Denmark. In the randomization process patients are stratified according to NIHSS (0-17 or > 17) and age (18-65 or > 66)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual blood pressure management arm (Experimental): During the EVT procedure(in general anesthesia), mean arterial blood pressure (MABP) during is targeted to remain within +/- 10 % of a reference value using vasoactive drugs and/or fluids
  Interventions: Procedure: Individualized blood pressure management
- Standard blood pressure management arm (Active Comparator): During the EVT procedure(in general anesthesia), mean arterial blood pressure (MABP) during is targeted to remain within a fixed range of 70-90 mmHg
  Interventions: Procedure: Standard blood pressure management

INTERVENTIONS:
Procedure: Individualized blood pressure management — During the EVT procedure, mean arterial blood pressure (MABP) is targeted to remain within +/- 10 % of a reference value using vasoactive drugs and/or fluids
  Arms: Individual blood pressure management arm
Procedure: Standard blood pressure management — During the EVT procedure, mean arterial blood pressure (MABP) is targeted to remain within a fixed range of 70-90 mmHg
  Arms: Standard blood pressure management arm

SUMMARY:
The ideal blood pressure management strategy during endovascular therapy (EVT) for acute ischemic stroke has not been defined. The aim of this pilot randomized clinical trial is to determine whether randomization to a standard versus individual blood pressure management strategy during the EVT procedure is feasible.

DETAILED DESCRIPTION:
Acute ischemic stroke (AIS) is a leading cause of death and long-term disability in the Western world. Catheter-based removal of blood clots (endovascular therapy-EVT) is now the standard of care for AIS caused by large vessel occlusions in the brain. The level of blood pressure during the procedure appears to influence outcome. However, optimal blood pressure management strategy has not been determined. Current blood pressure management strategy during EVT typically aims to maintain blood pressure above or within predefined fixed targets and is based on observational data and expert consensus rather than on high-quality randomized evidence. Should blood pressure during removal of the occlusion be managed according to the patient's individual blood pressure level or according to predefined fixed blood pressure targets? The primary aim of this pilot trial is to determine whether randomization to a procedure strategy targeting a predefined mean arterial blood pressure (MABP) of 70-90 mmHg versus an individual strategy targeting ± 10 % of a MABP reference value is feasible. Secondary aims are to test recruitability and to detect challenges or obstacles that would call for changes in the study design.

ELIGIBILITY:
Inclusion Criteria:

* Large vessel occlusion in anterior circulation in patients deemed treatable with EVT.
* Living independently (mRS < 2) before stroke.
* EVT procedure feasible within 24 hours of symptom onset.

Exclusion Criteria:

* Contra-indication/allergy to contrast agents, vasopressor agents or anaesthetics.
* Pregnancy.
* Medical condition where blood pressure targeting will be problematic (aorta dissection, etc).
* Participation in another trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-01-16 (Actual); Study Completion 2022-01-16 (Actual)

PRIMARY OUTCOMES:
3-month Modified Rankin Score (mRS). The mRS is a functional outcome score rankin from 0(best outcome) to 6 (death) | Assessed up to 3 months after endovascular treatment
  Functional outcome measure

SECONDARY OUTCOMES:
Recruitment rate (percentage) | Assessed up 3 months after endovascular treatment
  Percentage of admitted patients scheduled for EVT who is enrolled in the study
Adherence to mean arterial blood pressure targets. Specifically, to determine the percentage of time outside the target treatment range | Assessed 3 months after endovascular treatment
  ...Percentage of time outside the blood pressure targets
Data completeness (percentage) | Assessed up to 3 months after endovascular treatment
  Percentage of complete patient data study records
Degree of reperfusion | Assessed up to 3 months after endovascular treatment
  Thrombolysis in Cerebral Infarction Score (TICI) score. The TICI score is a grading scale for angiographic outcomes rankin from 0 (no perfusion) to 3(complete perfusion)

OTHER OUTCOMES:
Criteria for continuation to the definitive trial | Assessed up to 3 months after endovascular treatment
  The two arms are distinguishable on 3-month mRS with a trend statistical significant p-value below 0.1 or all of the following:
  * Drop out rate is less than 10%
  * Data completion is above 90%
  * (A cumulated duration of 10 minutes outside the MABP targets is allowed) Additional cumulated time outside the respective MABP target range is on average less than 8% of the duration of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mads Rasmussen, MD, PhD, Principal Investigator — Department of Anesthesia, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
This is a pilot study and the data may be made available to other researchers upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data may be shared after publication of main study results within a period of 5 years after publication
Access Criteria: No criteria